CLINICAL TRIAL: NCT00971061
Title: Ahmed Glaucoma Valve and Single-Plate Molteno Implants in Treatment of Refractory Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanak Eye Surgery Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1465087
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Refractory Glaucoma
Keywords: Ahmed valve; single-plate Molteno implant; refractory glaucoma; surgical treatment
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSPI (Experimental): Molteno single-plate implant
  Interventions: Device: Molteno single-plate implant (MSPI)
- AVI (Active Comparator): Ahmed valve implant
  Interventions: Device: Ahmed valve implant

INTERVENTIONS:
Device: Ahmed valve implant — 184 mm2 surface area Ahmed Glaucoma Valve (AGV Model FP7; New World Medical Inc., Rancho Cucamonga, California, USA)
  Arms: AVI
Device: Molteno single-plate implant (MSPI) — 134 mm2 surface area single-plate Molteno implant (Molteno Ophthalmic Limited, Dunedin, New Zealand)
  Arms: MSPI

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of the Ahmed valve implant (AVI) and the Molteno single-plate implant (MSPI) in eyes with refractory glaucoma during a follow-up period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* refractory glaucoma, defined as uncontrolled IOP despite maximal anti-glaucoma medication, previously failed nonseton surgical treatment, or a combination thereof.

Exclusion Criteria:

* age less than 40 years
* a visual acuity of no light perception
* lens opacity
* elevated IOP associated with silicone oil previous glaucoma drainage device implantation in the same eye
* previous cyclodestructive treatment
* increased risk of endophthalmitis posterior segment disorders
* pre-existing ocular comorbidities.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-01; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Intra Ocular pressure (IOP) | Month 24

SECONDARY OUTCOMES:
Intra Ocular pressure (IOP) | day 1,week 1, and months 1, 3, 6, 9, 12 and 18
Changes in visual acuity | day 1,week 1, and months 1, 3, 6, 9, 12, 18, and 24.
Number of anti-glaucoma medications | week 1, and months 1, 3, 6, 9, 12, 18, and 24
Mean deviation of visual field, | week 1, and months 1, 3, 6, 9, 12, 18, and 24
Rate of intra- and postoperative complications | week 1, and months 1, 3, 6, 9, 12, 18, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Nader Nassiri, MD, Principal Investigator — Assistant Professor, Department of Ophthalmology, Imam Hussein Medical Center, Shaheed Beheshti University of Medical Sciences, Tehran, Iran; Nariman Nassiri, MD, Principal Investigator — Medical Researcher, Vanak Eye Surgery Center, Tehran, Iran; Ghazal Kamali, MD, Principal Investigator — 4th-year Resident, Department of Ophthalmology, Imam Hussein Medical Center, Shaheed Beheshti University of Medical Sciences, Tehran, Iran
Locations (1):
- Vanak Eye Surgery Center, Tehran, Tehran Province, Iran